CLINICAL TRIAL: NCT04912115
Title: A Multi-Center, Phase II, Randomized, Double-Blind, Prospective, Active Placebo- Controlled Trial of Sub-Anesthetic Intravenous Infusion of Ketamine to Treat Levodopa- Induced Dyskinesia in Subjects With Parkinson's Disease
Brief Title: Randomized, Double-Blind, Active Placebo-Controlled Study of Ketamine to Treat Levodopa-Induced Dyskinesia
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Seeking Pivotal study initiation
Sponsor: PharmaTher Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-001
Record Dates: First submitted 2021-05-25; First posted 2021-06-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations
MeSH Terms: conditions — Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Ketamine will be administered as intravenous infusions with infusion rates ranging from 0.1 mg/kg/hr to 0.30 mg/kg/hr. To maintain blinding, both active and placebo will be infused at similar infusion rates (mL/hr).
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Midazolam will be administered as intravenous infusions with infusion rates ranging from 0.009 mg/kg/hr to 0.027 mg/kg/hr. To maintain blinding, both active and placebo will be infused at similar infusion rates (mL/hr).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Ketamine is an FDA-approved N-methyl-D-aspartate (NMDA) receptor-modulating drug pharmacologically classified as an NMDA receptor antagonist (also noted to be a weak opioid receptor agonist).
  Arms: Ketamine
Drug: Midazolam — Midazolam is a benzodiazepine used for anesthesia, procedural sedation, trouble sleeping, and severe agitation.
  Arms: Midazolam

SUMMARY:
A Multi-Center, Phase II, Randomized, Double-Blind, Prospective, Active Placebo-Controlled Trial of Sub-Anesthetic Intravenous Infusion of Ketamine to Treat Levodopa-Induced Dyskinesia in Subjects with Parkinson's Disease.

DETAILED DESCRIPTION:
This Phase II trial is a prospective, double-blind, randomized, parallel trial-design with two arms. Subjects will be randomized to treatment with the investigational product (ketamine) or an active control (midazolam). The active control causes mild sedation and is employed to minimize unmasking of the test article.

The study is an out-patient study. However, infusion days and days involving prolonged assessments are expected to require the subject to be onsite. Subjects will return to the site for safety and efficacy evaluations. On Day 1, PK samples will be collected near the end of Infusion 1 and post-infusion to evaluate near-steady-state blood levels in all subjects. Intensive PK sampling will be conducted in all subjects prior to, during, and a few hours after Infusion 2 (Day 5 ± 2).

The primary objective of the study is to evaluate the effects of low-dose intravenous infusion of ketamine on levodopa-induced dyskinesia (LID) in patients with Parkinson's disease. All patients included in the study should meet the inclusion criteria. Half of the participants will receive ketamine, while the other half will receive active placebo (Midazolam). All participants will be assigned to either the active group or the control group randomly. During the clinical trial, both investigators and patients are double-blind except serious adverse events occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Parkinson's Disease as defined by the UK Parkinson's Disease Society Brain Bank Criteria
2. Signed a current IEC approved informed consent form
3. Male or female patients between ages 30-85 years
4. At least three years of prior treatment with levodopa of at least 400 mg daily subject to a maximum of 8 divided doses per day (excluding bedtime and nighttime)
5. Waking day dyskinesia of > 25% determined as a score of ≥2 as per Question 4.1 on the UPDRS
6. Ambulatory or ambulatory-aided (e.g., walker or cane) and able to complete study assessments
7. Have been on stable doses of all anti-Parkinson's medications for 30 days prior to entry into the study, including a levodopa preparation administered not less than three times daily, and be willing to remain on the same doses of medications throughout the course of the study
8. Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and the patient must be willing to continue the same doses and regimens during study participation.
9. The subject/caregiver must demonstrate the ability to complete an accurate home diary based on training and evaluation (visit 2)
10. Subjects must have available a responsible adult caregiver/companion who will drive the subject home following infusions
11. Female subjects not of childbearing potential
12. Male subjects, regardless of their fertility status, with nonpregnant women of childbearing potential (WOCBP) partners must agree to either remain abstinent (if this is their preferred and usual lifestyle) or use a highly effective (less than 1% failure rate) method of contraception (such as combination oral contraceptives, implanted contraceptives, or intrauterine devices) or effective method of contraception (such as diaphragms with spermicide or cervical sponges) for the duration of the study and until their plasma concentrations are below the level that could result in a relevant potential exposure to a possible fetus, predicted to be 90 days following the last dose of study drug

Exclusion Criteria:

1. Diagnosis of an atypical or secondary Parkinsonian syndrome
2. Lack of documented response to levodopa
3. Hoehn and Yahr stage of 5
4. Known prior exposure to ketamine or other NMDA inhibitors within the last 30 days
5. History of neurosurgical intervention related to PD (e.g., deep brain stimulation)
6. History of seizures within two years prior to screening
7. History of transient ischemic attacks or stroke within two years prior to screening
8. History of intracerebral hemorrhage due to hypertension.
9. History of clinically significant arrhythmia or unstable angina within the past five years
10. History of myocardial infarction within 2 years prior to screening
11. History of NYHA Class 3 or 4 heart failure within 2 years prior to screening
12. Aneurysmal vascular disease (e.g., intracranial, thoracic or abdominal aorta)
13. History of hypertensive encephalopathy

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Unified Dyskinesia Rating Scale (UDysRS) total score from Baseline to Week 8. | 8 weeks
  The change from baseline to week 8 of treatment in the sum of the items comprising the Unified Dyskinesia Rating Scale (UDysRS). The Unified Dyskinesia Rating Scale (UDysRS) is administered to assess dyskinesia. The scoring range is 0-104, where higher score means more dyskinesia.

SECONDARY OUTCOMES:
Change in total daily OFF times as assessed by subject completed 24-hour diaries, from Baseline to Week 8. | 8 weeks
  Change in daily "OFF"-time as assessed with patient diaries from run-in to week 8. This is a self administered diary where patients assess their motor state every half hour during 24 hours.
Change in the UPDRS total score of part III (motor) and sum score of Questions 4.1 and 4.2 (dyskinesia) in part IV from Baseline to Week 8. | 8 weeks
  Change in MDS-UPDRS sum score of part III (Motor Examination) from baseline to week 8. Minimum value is 0 and maximum value is 124. Higher score mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — PharmaTher Inc.
Locations (7):
- United States (7):
  - Investigative Site #7, Tucson, Arizona
  - Investigative Site #2, Chula Vista, California
  - Investigative Site #1, Fountain Valley, California
  - Investigative Site #3, Miami, Florida
  - Investigative Site #6, Miami, Florida
  - Investigative Site #5, Rolling Meadows, Illinois
  - Investigative Site #4, Plymouth, Michigan